CLINICAL TRIAL: NCT06564142
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study of Povetacicept in Adults With Immunoglobulin A Nephropathy (RAINIER)
Brief Title: Evaluation of Efficacy of Povetacicept in Adults With Immunoglobulin A Nephropathy (IgAN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alpine Immune Sciences Inc, A Subsidiary of Vertex (Industry)
Responsible Party: Sponsor
Organization: Alpine Immune Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX24-AIS-D08; 2024-514135-17-00 (Other: EU CT number)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Immunoglobulin A Nephropathy
Keywords: IgAN; Berger's disease; glomerulonephritis; IgA nephropathy; ALPN-303; BAFF; BLyS; APRIL
MeSH Terms: conditions — Glomerulonephritis, IGA; Glomerulonephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Povetacicept (Experimental): Participants will be randomized to receive Povetacicept.
  Interventions: Drug: Povetacicept
- Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to Povetacicept.
  Interventions: Drug: Placebo (matched to Povetacicept)

INTERVENTIONS:
Drug: Povetacicept — Subcutaneous injection administration.
  Other Names: ALPN-303
  Arms: Povetacicept
Drug: Placebo (matched to Povetacicept) — Placebo matched to Povetacicept subcutaneous injection administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of povetacicept in adult participants compared with placebo in reducing proteinuria and preserving renal function.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed IgAN, with biopsy confirmation
* 24-hr proteinuria excretion ≥1.0 g/day or 24-hour uPCR ≥0.75 g/g
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73m^2
* Stable angiotensin converting enzyme inhibitor (ACEi) or angiotensin II receptor blocker (ARBs) as per protocol specification

Key Exclusion Criteria:

* Have received any immunosuppressive treatment or procedures (including corticosteroids, oral immunosuppressive agents, B cell or plasma cell targeted therapies, complement targeted therapies, herbal medicines per protocol, and tonsillectomy) within a wash-out period per protocol
* Rapidly progressive glomerulonephritis with eGFR reduction >50% within 12 weeks of the start of screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in 24-hour Urine Protein to Creatinine Ratio (uPCR) at Week 36 | From Baseline at Week 36
Total Estimated Glomerular Filtration Rate (eGFR) Slope Through Week 104 | From Baseline Through Week 104

SECONDARY OUTCOMES:
Change from Baseline in Serum Gd-IgA1 at Week 36 | From Baseline at Week 36
Proportion of Participants to Achieve Hematuria Resolution at Week 36 (Among Participants With Hematuria at Baseline) | From Baseline at Week 36
Change From Baseline in eGFR at Week 104 | From Baseline at Week 104
Time to Kidney Disease Progression Through Week 104 | From Baseline Through Week 104
  Kidney disease progression defined as greater than or equal to (≥) 30% decline in eGFR, end stage kidney disease, or non-accidental death

CONTACTS AND LOCATIONS:
Locations (318):
- United States (77):
  - Apogee Clinical Research, LLC, Huntsville, Alabama
  - Arizona Kidney Disease and Hypertension Center - Thomas Office, Phoenix, Arizona
  - Arizona Kidney Disease and Hypertension Center - Tuscon, Tucson, Arizona
  - West Coast Kidney, Fremont, California
  - The Medical Research Group, Inc. (FRENOVA), Fresno, California
  - CARE Institute - Carabello Kidney, Los Angeles, California
  - Providence Medical Foundation - Orange, Orange, California
  - National Nephrology Alliance Research, Riverside, California
  - UC Davis Health, Sacramento, California
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Western Nephrology, Arvada, Colorado
  - Colorado Kidney Care, Denver, Colorado
  - Nephrology Associates Delaware Kidney (FRENOVA), Newark, Delaware
  - South Florida Nephrology Group PA, Research Div., Coral Springs, Florida
  - Dolphin Medical Research, Doral, Florida
  - Nephrology Associates of Central Florida, Hollywood, Florida
  - Tectum Medical Research, LLC, Hollywood, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Florida Kidney Physicians - Melbourne, Melbourne, Florida
  - Med-Care Research, Miami, Florida
  - Professional Research Center, Miami, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - On Health Research Center, Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - BioResearch Partner, Pembroke Pines, Florida
  - D&H Pompano Research Center, Pompano Beach, Florida
  - Cordova Research Institute, LLC, Sweetwater, Florida
  - SciMerge Clinical Research, Atlanta, Georgia
  - Georgia Nephrology - Lawrenceville, Lawrenceville, Georgia
  - Randomize Now - Midtown, Newnan, Georgia
  - Care Institute - Chubbuck, ID, Chubbuck, Idaho
  - Care Institute - Idaho Falls, Idaho Falls, Idaho
  - CARE - Boise Kidney Institute, Meridian, Idaho
  - Bioluminux Clinical Research, Naperville, Illinois
  - Rockford Nephrology Associates, Rockford, Illinois
  - Nephrology Associates of Northern Illinois and Indiana (NANI), Indianapolis, Indiana
  - Nephrology Physicians LLC, Mishawaka, Indiana
  - Nephrology Associates of Kentuckiana, Louisville, Kentucky
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Velocity Clinical Research - Metairie, Metairie, Louisiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - St. Clair Nephrology Research, Shelby, Michigan
  - InterMed Consultants / DaVita Clinical Research, Edina, Edina, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Nephrology and Hypertension Associates, LTD, Tupelo, Mississippi
  - Washington University in St. Louis, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - DaVita Clinical Research Nevada - Las Vegas, Las Vegas, Nevada
  - Bioluminux Clinical Research New Jersey, Hamilton, New Jersey
  - New Jersey Kidney Care, LLC (FRENOVA), Jersey City, New Jersey
  - Renal Medicine Associates, Albuquerque, New Mexico
  - New York Nephrology Vasculitis and Glomerular Center, Albany, New York
  - Queens Hospital Center, Jamaica, New York
  - The Rogosin Institute, New York, New York
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Nephrology Associates Inc, East Providence, Rhode Island
  - Hypertension & Nephrology Inc., Providence, Rhode Island
  - South Carolina Clinical Research, LLC, Orangeburg, South Carolina
  - Knoxville Kidney Center (KKC), PLLC, Knoxville, Tennessee
  - Velocity Clinical Research, Abilene, Texas
  - Introscience Research LLC, Bellaire, Texas
  - Dallas Renal Group, Dallas, Texas
  - Renal Disease Research Institute - Dallas, Dallas, Texas
  - Davita Clinical Research - El Paso, El Paso, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Houston Medical Research Institute, LLC (FRENOVA), Houston, Texas
  - R & H Clinical Research, Katy, Texas
  - North Texas Kidney Disease Associates, Lewisville, Texas
  - P&I Clinical Research, LLC, Lufkin, Texas
  - Renal Specialists of Houston, Pasadena, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
  - Virginia Nephrology Group, Fairfax, Virginia
  - Kidney and Hypertension Specialist PLLC, Manassas, Virginia
- Australia (17):
  - Grampians Health Ballarat, Ballarat
  - Bendigo Hospital, Bendigo
  - Sunshine Coast University Hospital, Birtinya
  - Core Research Group Pty Ltd, Brisbane
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Health, Clayton
  - Concord Repatriation General Hospital, Concord
  - Canberra Hospital, Garran
  - Renal Research Gosford, Gosford
  - Austin Hospital, Heidelberg
  - Western Health (Sunshine Hospital), Melbourne
  - Fiona Stanley Hospital, Murdoch
  - John Hunter Hospital, Newcastle
  - Sir Charles Gairdner Hospital, Perth
  - Melbourne Renal Research, Reservoir
  - Gold Coast University Clinical Trials Unit, Southport
  - Princess Alexandra Hospital, Woolloongabba
- Austria (5):
  - LKH Feldkirch, Feldkirch
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Medizinische Universitaet Wien, Vienna
  - Klinikum Wels- Grieskirchen, Wels-Grieskirchen
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (18):
  - Centro de Pesquisa Clinica do Coracao, Aracaju
  - Freire Pesquisa Clinica, Belo Horizonte
  - Hospital Evangelico de Belo Horizonte, Belo Horizonte
  - Associacao Ampara a Saude, Brasília
  - HU Hospital Walter Cantidio, Fortaleza
  - UFG Hospital de Clinicas da Universidad Federal de Golas, Goiânia
  - Hospital de Caridade de Ijui, Ijuí
  - Fundacao Pro-Rim Santa Catarina, Joinville
  - Centro Mineiro de Pesquisa, Juiz de Fora
  - Hospital das Clinicas Riberao Preto, Monte Alegre
  - Hospital das Clinicas da Universidade Federal de Pernambuco (UFPE), Recife
  - Hospital Universitario Pedro Ernesto - UERJ, Rio de Janeiro
  - Clinica Senhor do Bonfim, Salvador
  - Universidade Federal da Bahia, Salvador
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Hospital do Rim Fundacao Oswaldo Ramos, São Paulo
  - Hospital Nove de Julho - DASA, São Paulo
  - A2z Clinical Centro Avancedo de Pesquisa Clinica, Valinhos
- St. Josephs Healthcare - Hamilton, Hamilton, Canada
- China (45):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University First Hos, Beijing
  - Cangzhou People's Hospital, Cangzhou
  - The Second Norman Bethune Hospital of Jilin University, Changchun
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Sichuan People s Hospital, Chengdu
  - Bishan Hospital of Chongqing, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Dongguan People s Hospital, Dongguan
  - The First People's Hospital of Foshan, Foshan
  - Fuyang People's Hospital, Fuyang
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Third Affiliated Hospital of Southern Medical University, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Affiliated Hospital of Guilin Medical University, Guilin
  - Guizhou Provincial People's Hospital, Guiyang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan
  - The Second Hospital of Shandong University, Jinan
  - Linyi People's Hospital, Linyi
  - The First Affiliate Hospital of Henan University of Science and Technology, Luoyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Hospital of Nantong University, Nantong
  - Ningbo No.2 Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - The First Affiliated Hospital of Xian JiaoTong University, Shaanxi
  - Shanghai General Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - Taian City Central Hospital, Taian
  - Second Hospital of Shanxi Medical University, Taiyuan
  - The Second Hospital of Tianjin Medical University, Tianjin
  - Wuxi People s Hospital, Wuxi
  - Xuancheng People s Hospital, Xuancheng
  - Yancheng No. 1 People's Hospital, Yancheng
  - Affiliated Hospital Yangzhou University, Yangzhou
  - Yantai YuHuangDing Hospital, Yantai
  - Yichang central people Hos, Yichang
  - General Hospital of Ningxia Medical University, Yinchuan
- Croatia (3):
  - Clinical Hospital Dubrava, Zagreb
  - Clinical Hospital Merkur, Zagreb
  - Polyclinic Somed, Zagreb
- Czechia (3):
  - Fakultni Nemocnice Brno, Brno
  - Vseobecna fakultni nemocnice v Praze, New Town
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Center for Cancer and Organ Diseases - Rigshospitalet - Hornum Mads, Copenhagen
  - Hillerod Hospital, Hillerød
  - Sygehus Lillebaelt - Kolding, Kolding
- Estonia (2):
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- Tampere University Hospital, Tampere, Finland
- France (9):
  - Groupe Hospitalier Pellegrin, CHU De Bordeaux, Bordeaux
  - Hopitaux Universitaires Henri Mondor, Créteil
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - AP-HM - Hopital de La Conception, Marseille
  - CHU de Nantes - Hotel-Dieu, Nantes
  - Hopital Necker - Enfants Malades, Paris
  - Université Paris-Descartes / Hôpital Européen Georges Pompidou, Paris
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Centre Hospitalier de Valencienes, Valenciennes
- Germany (5):
  - Medizinische Klinik II, Aachen
  - Charite Universitaetsnedizin Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Klinikum St Georg, Leipzig
  - Universitaetsklinikum Leipzig, Leipzig
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Prince Wales Hospital, Shatin
  - Tung Wah Hospital, Sheung Wan
- Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs, Hungary
- Ireland (4):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Waterford, Waterford
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Rabin Medical Center, Petah Tivka
  - Sheba Medical Center, Tel Litwinsky
  - Shamir Medical Center, Ẕerifin
- Italy (5):
  - Azienda Ospedaliera Universitaria Consorziale - policlinicio Bari, Bari
  - Ospedale Policlinico San Martino IRCCS, Genova
  - AOU Policlinico di Modena, Modena
  - Istituti Clinici Scientifici Maugeri-IRCCS Pavia, Pavia
  - Fondazione Policlinico Universitario A. Gemelli, Rome
- Japan (29):
  - Fujita Health University Hos, Aichi
  - Hyogo Amagasaki Gen Med Ctr, Amagasaki
  - Fukuoka University Hospital, Fukuoka
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Nihon University Itabashi Hospital, Itabashi-ku
  - Kanazawa Medical Uni Hospital, Kahoku
  - Kanazawa University Hospital, Kanazawa
  - Nara Med University Hos, Kashihara
  - Kasugai Municipal Hospital, Kasugai
  - Okayama University Hospital, Kita-ku
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Kobe University Hospital, Kobe
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - University of Miyazaki Hos, Miyazaki
  - Osaka City General Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Sapporo City General Hospital, Sapporo
  - Tohoku University Tohoku University Hospital, Sendai
  - Juntendo Hospital Affiliated to Juntendo University School of Medicine, Tokyo
  - Juntendo University Nerima Hospital, Tokyo
  - The Jikei Uni Daisan Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - Tokyo Med University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - YUUAI Medical Center, Tomigusuku
  - Toyama Prefectural Central Hospital, Toyama
  - Juntendo Uni Urayasu Hospital, Urayasu-shi
- Latvia (2):
  - Paula Stradina Clinical University Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences (LSMU) Kauno klinikos, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Arke SMO SA de CV, Veracruz, Mexico
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - UMC St. Radboud, Nijmegen
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital - Ulleval Hospital, Oslo
- Poland (5):
  - SCM Sp. Z o.o, Krakow
  - Klinika Nefrologii, Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodzkie
  - Uniwersytecki Szpital Kliniczny nr 2 PUM w Szczecinie, Szczecin
  - Panstwowy Instytut Medyczny MSWiA - Klinika Chorob Wewnetrznych, Nefrologii i Transplantologii, Warsaw
  - Velocity Zamosc, Zamość
- Saudi Arabia (2):
  - King Fahad Specialist Hospital, Dammam, Dammam
  - King Saud University, King Saud University Medical City, Riyadh
- South Korea (22):
  - Hallym University Sacred Heart Hospital, Anyang
  - Seoul National University Hospital, Cheonan
  - Soon Chun Hyang University Cheonan Hospital, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Hallym University Chuncheon Sacred Heart Hospital, Gangwon-do
  - Wonju Severance Christian Hospital, Gangwon-do
  - NHIS Ilsan Hospital, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Medical Center (KUMC)-Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong (KUIMS), Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yongin Severance Hospital, Yongin-si
- Spain (12):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitatio Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari Arnau de Vilanova - Lleida, Lleida
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Sweden (5):
  - Nephrology Clinic, Danderyd University Hospital, Danderyd
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital Huddinge, Huddinge
  - Linkoping University Hospital, Linköping
  - Uppsala University Hospital, Uppsala
- Taiwan (5):
  - Shuang Ho Hospital, New Taipei City
  - Tungs' Taichung Metroharbour Hospital, Taichung
  - National Taiwan University Hospital (NTUH), Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital (TP-VGH), Taipei
- Turkey (Türkiye) (3):
  - Hacettepe University Hospital, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Kocaeli University Medical School, Kocaeli
- United Kingdom (17):
  - Belfast Health and Social Care Trust, Belfast
  - FutureMeds - Soho Road Health Centre, Birmingham
  - Southmead Hospital, Bristol
  - Cambridge University - Addenbrooke's Hospital, Cambridge
  - FutureMeds - CPS Research, Glasgow
  - Queen Elizabeth University Hospital - Glasgow, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Leicester General Hospital, Leicester
  - Barts Health NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - King's College Hospital, London
  - St Pancras Clinical Research, London
  - University of Manchester, Manchester Royal Infirmary, Manchester
  - FutureMeds Newcastle, Newcastle upon Tyne
  - FutureMeds Tesside, Stockton-on-Tees
  - FutureMeds Liverpool, Wirral (Liverpool)
  - Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/